CLINICAL TRIAL: NCT03264638
Title: A Clinical and Biological Research of Combined Chinese and Western Medicine in the Treatment of Polycystic Ovary Syndrome
Brief Title: A Clinical and Biological Research of Combined Chinese and Western Medicine in the Treatment of PCOS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aijun Sun (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Tang-Du Hospital (Other)
Responsible Party: Sponsor-Investigator, Aijun Sun, Principal Investigator, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCOS201708
Record Dates: First submitted 2017-08-13; First posted 2017-08-29 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: PCOS
Keywords: PCOS; Dingkundan; Diane-35
MeSH Terms: interventions — Cyproterone acetate, ethinyl estradiol drug combination

STUDY DESIGN:
Intervention Model Description: One third of participanta will receive Dingkun Dan Pills, one third of participanta will receive Diane-35 Pills, and the another third will receive Dingkun Dan pills and Diane-35 in combination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dingkundan (Experimental): Dingkundan 7g capsule by mouth, twice daily, beginning on Day 5 of menstrual cycle for 21 consecutive days followed by a 7-day interval without medication; for three cycles
  Interventions: Drug: Dingkundan
- Dingkundan & Diane-35 (Experimental): Dingkundan 7g capsule by mouth, twice daily, and Diane-35 one pill by mouth, once daily, beginning on Day 5 of menstrual cycle for 21 consecutive days followed by a 7-day interval without medication; for three cycles
  Interventions: Drug: Dingkundan & Diane-35
- Diane-35 (Active Comparator): Diane-35 one pill by mouth,once daily, beginning on Day 5 of menstrual cycle for 21 consecutive days followed by a 7-day interval without medication; for three cycles
  Interventions: Drug: Diane-35

INTERVENTIONS:
Drug: Dingkundan — Dingkundan 7g capsule by mouth, twice daily, beginning on Day 5 of menstrual cycle for 21 consecutive days followed by a 7-day interval without medication; for three cycles
  Other Names: A
  Arms: Dingkundan
Drug: Dingkundan & Diane-35 — Dingkundan 7g capsule by mouth, twice daily, and Diane-35 one pill by mouth, once daily, beginning on Day 5 of menstrual cycle for 21 consecutive days followed by a 7-day interval without medication; for three cycles
  Other Names: A&B
  Arms: Dingkundan & Diane-35
Drug: Diane-35 — Diane-35 one pill by mouth,once daily, beginning on Day 5 of menstrual cycle for 21 consecutive days followed by a 7-day interval without medication; for three cycles
  Other Names: B
  Arms: Diane-35

SUMMARY:
This study evaluates the effects and biological mechanisms of Dingkundan，Diane-35 and the combination of Dingkundan and Diane-35 in the treatment of polycystic syndrome(PCOS) in adults women. One third of participants will receive Dingkundan capsules, one third of participants will receive Diane-35 Pills, and the another third will receive Dingkundan capsules and Diane-35 in combination.

DETAILED DESCRIPTION:
Dingkundan,Diane-35 each ameliorate PCOS, but they do so by different mechanisms. We generally treat PCOS patients without immediate fertility requirement by short-acting contraceptives,Diane-35 is one of the most commonly used drugs.

Dingkundan consists of multiple chinese herbs including ginseng,Panax notoginseng,deer antlers,Carthamus tinctorius L.,Radix Paeoniae Alba,prepared Radix Rehmanniae,Angelica etc., which gains widespread application in the treatment of gynecological diseases. Based on the characteristics above, we try to explore its clinical application value in PCOS and its biological mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a female between the age of 18 and 40.
* Subject diagnosed as PCOS by the 2003 Rotterdam criteria.
* Subject provides written informed consent.

Exclusion Criteria:

* Subject has other endocrine diseases,such as adrenal hyperplasias or tumor, androgen-secreting tumours, Cushing's syndrome,thyroid diseases and hyperprolactinemia.
* Subject has received related medical or surgical treatment in the past 3 months.
* Subject suffered from substance abuse or dependence(such as alcohol or drugs);
* Subject is a heavy smoker(reaching or more than 20 cigarettes a day).
* Subject is pregnant or lactating or within 1 year after delivery.
* Subject has a severe systemic disease, such as cardiovascular system
* Subject has a history of malignancy or radiotherapy.
* Subject has an allergic history to the drugs used in the study.
* Subject has mental disorder incapable of elementary cooperations.
* Subject has participated in other clinical researches of medicine within 3 month prior to randomization.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 315 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
symptoms | 5 minutes
  PCOS symptoms
sex hormone levels changes | 5 minutes
  sex hormone levels changes

SECONDARY OUTCOMES:
lipid metabolism | 5 minutes
  blood lipid profile
metabolites figure spectrum | 5 minutes
  metabolites figure spectrum to undermine the mechanism of Dingkundan and Diane-35 in the treatment of PCOS
Fasting insulin | 5 minutes
  Fasting insulin
glycosylated hemoglobin | 5 minutes
  glycosylated hemoglobin
fasting blood glucose | 5 minutes
  fasting blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Aijun Sun, MD, Principal Investigator — Peking Union Medical College Hospital,Peking Union Medical College, Chinese Academy of Medicine Sciences
Locations (1):
- Lei Li, Beijing, China/Beiing, China

IPD SHARING:
Plan to Share IPD: Yes
Network platform, and the website will be attached later.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Within 2 months after the trial complete
Access Criteria: Data access requests will be reviewed by an external independent review panel.Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS consensus workshop group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS). Hum Reprod. 2004 Jan;19(1):41-7. doi: 10.1093/humrep/deh098. PMID 14688154
- [Background] Amiri M, Ramezani Tehrani F, Nahidi F, Kabir A, Azizi F, Carmina E. Effects of oral contraceptives on metabolic profile in women with polycystic ovary syndrome: A meta-analysis comparing products containing cyproterone acetate with third generation progestins. Metabolism. 2017 Aug;73:22-35. doi: 10.1016/j.metabol.2017.05.001. Epub 2017 May 10. PMID 28732568
- [Derived] Ding X, Deng Y, Wang Y, Xue W, Zhu S, Ma X, Ma R, Sun A. Serum metabolomic profiling reveals potential biomarkers in assessing the management of women with polycystic ovary syndrome: a randomized controlled trial. Chin Med J (Engl). 2022 Jan 5;135(1):79-85. doi: 10.1097/CM9.0000000000001705. PMID 34873082
- [Derived] Deng Y, Wang YF, Zhu SY, Ma X, Xue W, Ma RL, Sun AJ. Is There An Advantage of Using Dingkun Pill () alone or in Combination with Diane-35 for Management of Polycystic Ovary Syndrome? A Randomized Controlled Trial. Chin J Integr Med. 2020 Dec;26(12):883-889. doi: 10.1007/s11655-020-3097-4. Epub 2020 Sep 11. PMID 32915426
- [Derived] Deng Y, Xue W, Wang YF, Liu XH, Zhu SY, Ma X, Zuo HL, Jiang JF, Zheng TP, Sun AJ. Insulin Resistance in Polycystic Ovary Syndrome Improved by Chinese Medicine Dingkun Pill (): A Randomized Controlled Clinical Trial. Chin J Integr Med. 2019 Apr;25(4):246-251. doi: 10.1007/s11655-018-2947-1. Epub 2019 Jun 25. PMID 31236888
- See also: Diane can be used to ameliorate acne in PCOS patients — http://www.newhealthguide.org/Diane-Pills.html